CLINICAL TRIAL: NCT06479915
Title: Access the Influence of Oral Microbiota in the Onset and Evolution of Stroke, With Focus on Cerebral Microbleeds
Brief Title: Estimate the Relationship Between Oral Microbiota and Stroke
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Collaborators: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xiaojing Huang, Archiater, Fujian Medical University
Other Study IDs: SHFMU
Record Dates: First submitted 2024-06-19; First posted 2024-06-28 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Microbial Disease
Keywords: cnm; Streptococcus mutans; Cerebal microbleeds; Cerebral hemorrhage; Cerebral ischemia; cnm-positive streptococcus mutans
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage; Brain Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva;dental plaque
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Stroke: Small cerebral vessel disease
- healthy people: MRI showed no signs of small cerebral vessel disease

SUMMARY:
Oral bacteria constitute the second largest population of the human microbiome. Recent studies have identified their role in the development of systemic diseases, such as cardiovascular and cerebrovascular diseases. Streptococcus Mutans (SM) is considered the primary pathogen responsible for dental caries. Furthermore, in cases of oral inflammatory diseases, SM has been found to invade the bloodstream and disseminate, leading to systemic diseases. Against this backdrop, this study aims to investigate disparities in oral flora between stroke patients and healthy individuals by collecting saliva samples from both groups.

DETAILED DESCRIPTION:
Oral bacteria constitute the second largest population of the human microbiome. Recent studies have identified their role in the development of systemic diseases, such as cardiovascular and cerebrovascular diseases. Streptococcus Mutans (SM) is considered the primary pathogen responsible for dental caries. Furthermore, in cases of oral inflammatory diseases, SM has been found to invade the bloodstream and disseminate, leading to systemic diseases. Against this backdrop, this study aims to investigate disparities in oral flora between stroke patients and healthy individuals by collecting saliva samples from both groups. The objective of this study is to offer novel insights into the association between oral health and cerebrovascular disease occurrence while establishing a foundation for future research.

ELIGIBILITY:
Inclusion Criteria:

* 1. Microbleeding/damage or rupture of small blood vessels in the brain has been diagnosed within the past 365 days 2. Have done nuclear magnetic examination and can provide nuclear magnetic results

Exclusion Criteria:

* Have received antibiotic quality within the last three months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: small cerebral vessel disease
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Estimate the Relationship Between Oral Microbiota and Stroke | 2025.06
  Measure the diversity and abundance of oral bacteria in stroke patients,units:Number of bacterial species, bacterial counts (CFU/ml)
Correlation Between Oral Microbiota and Cerebral Microbleeds in Stroke | 2025.06
  Number and volume of microbleeds (measured in mm³)

CONTACTS AND LOCATIONS:
Overall Officials: XiaoJing Huang, Study Chair — School and Hospital of Stomatology,Fujian Medical University,fuzhou,Fujian Province,350002,China
Locations (2):
- China (2):
  - School and Hospital of stomatology,Fujian Medical University,Fuzhou,Fujian Province,350002,China, Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian